CLINICAL TRIAL: NCT03876626
Title: Using Smart Phone Technology to Support HIV Medication Refill Adherence in Virginia - Pilot Study
Brief Title: Using Smart Phone Technology to Support HIV Medication Refill Adherence in Virginia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Virginia Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21185
Record Dates: First submitted 2019-02-25; First posted 2019-03-15 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Hiv; Adherence, Medication
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provider Participants (Other): Employees who work with medication refills through the AIDS Drug Assistance Program at the Henrico Health Department will be invited to participate in the study as providers. Provider participants will receive access to a web based system that allows them to view information for their enrolled clients, securely message clients, and track medication refills. Providers will be asked to participate in a 30-day usability interview and a end-of-study assessment.
  Interventions: Other: PositiveLinks RX Portal
- Patient Participants (Other): Clients who receive medication refills through the AIDS Drug Assistance Program at the Henrico Health Department will be invited to participate in the study as patients. Patient participants will be provided access to a mobile app that allows them to track their mood, stress, and medication adherence, access an anonymous online community, securely message providers, and receive medication refill alerts
  Interventions: Other: PositiveLinks RX Mobile App

INTERVENTIONS:
Other: PositiveLinks RX Mobile App — A mobile app designed with tools to facilitate patient self-monitoring, patient-provider communication, medication refills, and social support.
  Arms: Patient Participants
Other: PositiveLinks RX Portal — An online portal that interacts with the mobile app to enable users to engage with participants though messaging and medication refill tracking.
  Arms: Provider Participants

SUMMARY:
The purpose of this study is to pilot a mobile health intervention, originally designed for HIV retention in care, for use in aiding patients with medication refills. The study will implement the PositiveLinks Rx app with the Henrico Health department. The study will assess user engagement and satisfaction with the app as well as preliminary impact on patient refill compliance.

DETAILED DESCRIPTION:
The study will enrolled provider and patient participants at the Henrico Health Department in Virginia who either receive or provide medication refills through the AIDS Drug Assistance Program (ADAP). Patient participants will be provided access to a mobile app that allows them to track their mood, stress, and medication adherence, access an anonymous online community, securely message providers, and receive medication refill alerts. Provider participants will be able to view the information entered by enrolled clients, securely message clients, and track medication refill processes. Study participants will be asked to provide feedback on usability, utility, impact, and effectiveness of the program. Additional assessments will evaluate for impact on medication refill adherence and patient-provider communication.

ELIGIBILITY:
Patient Inclusion Criteria:

* Currently picking up of receiving medications through ADAP from the Henrico Health Department; Able to read in English; Able to speak English; Able to sign informed consent

Provider Inclusion Criteria:

* Current Henrico Health Department employee working with the ADAP pharmacy; Able to read in English; Able to speak English; Able to sign informed consent

Exclusion Criteria:

* Severe cognitive impairment that interferes with a subjects ability to consent; non-English speaking; Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Change in Patient Medication Refill Compliance | Assessed at baseline and 6-months
  Primary variable analysis will include examination of patient medication refill compliance at baseline and at the 6-month follow-up to assess for any change in refill compliance.

SECONDARY OUTCOMES:
App Usability | 30-days after enrollment
  Assessed through the system usability scale (SUS), a validated ten item scale. Additional usability factors will be assessed through qualitative methods.
Participant Check-In Engagement | Assessed at 6-months
  Examining participant app engagement through assessment of check-in response rates
Participant Messaging Engagement | Assessed at 6-months
  Examining participant app engagement through assessment of messages sent and received
Participant Community Engagement | Assessed at 6-months
  Examining participant app engagement through assessment of community posts
Participant Feature Engagement | Assessed at 6-months
  Examining participant app engagement through assessment of page views
Change in Patient Refill Satisfaction | Assessed at baseline and 6-months
  Assessment of change in patient satisfaction with the refill process at their local health department. Utilizes a patient satisfaction with pharmaceutical services scale.
Change in Provider Communication | Assessed at baseline and 6-months
  Assessment of change in patient perception of provider (local health department staff) communication. Utilizes the Consultation and Relational Empathy (CARE) scale.
Program Alignment with Health Department Workflow | Assessed at 30-days and 6-months
  Assessing alignment with health department workflow through provider end-of-study and usability interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Henrico Health Department, Richmond, Virginia, United States